CLINICAL TRIAL: NCT07268573
Title: Acute Effects of Combined and Isolated Caffeine and Theanine Supplementation on Physical and Cognitive Performance in Competitive Athletes: A Randomized, Double-Blind, Placebo-Controlled Crossover Study
Brief Title: Effects of Caffeine and L-Theanine on Physical and Cognitive Performance in Trained Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulaş Can YILDIRIM (Other)
Responsible Party: Sponsor-Investigator, Ulaş Can YILDIRIM, Assoc. Prof., Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2025/337
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Performance; Physical Performance Enhancement; Caffeine and L-theanine Interaction
MeSH Terms: interventions — Caffeine; theanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Caffeine Supplementation (CAF) (Experimental): Participants receive 3 mg of anhydrous caffeine per kilogram of body weight, encapsulated in gelatin capsules identical in appearance to other conditions. Capsules are ingested with water 60 minutes before testing.
  Interventions: Dietary Supplement: Caffeine
- L-Theanine Supplementation (THE) (Experimental): Participants receive 200 mg of L-theanine (pure L-theanine powder, Orzax Pharmaceuticals, Istanbul, Turkey), encapsulated in gelatin capsules identical in appearance to other conditions. Capsules are ingested with water 60 minutes before testing.
  Interventions: Dietary Supplement: L-theanine
- Combined Caffeine and L-Theanine (COM) (Experimental): Participants receive a combination of 3 mg/kg anhydrous caffeine and 200 mg L-theanine, encapsulated together in identical gelatin capsules. Capsules are taken 60 minutes before testing to assess potential synergistic effects on physical and cognitive performance.
  Interventions: Dietary Supplement: Combined Caffeine and L-Theanine
- Placebo (CON) (Placebo Comparator): Participants receive placebo capsules filled with mannitol, a non-nutritive sugar alcohol with no known ergogenic properties. Capsules are identical in size, color, texture, and weight to the active supplement conditions and are ingested 60 minutes before testing.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — Participants receive 3 mg of anhydrous caffeine per kilogram of body weight, encapsulated in identical gelatin capsules (five in total). Capsules are taken orally with water 60 minutes before testing. The caffeine powder (98.5% purity, Oxford Vitality Health Co., UK) is administered once per experimental session, with at least 72 hours between conditions.
  Arms: Caffeine Supplementation (CAF)
Dietary Supplement: L-theanine — Participants receive a single 200 mg dose of L-theanine (Orzax Pharmaceuticals, Istanbul, Turkey; active ingredient manufactured in Germany) encapsulated in identical gelatin capsules. The supplement is ingested orally with water 60 minutes before testing. All testing sessions are separated by at least 72 hours.
  Arms: L-Theanine Supplementation (THE)
Dietary Supplement: Combined Caffeine and L-Theanine — Participants receive a combination of 3 mg/kg anhydrous caffeine and 200 mg L-theanine, encapsulated together in visually identical gelatin capsules. The mixture is taken orally with water 60 minutes before testing to assess potential synergistic effects on performance. Each participant completes all four supplementation conditions in randomized order, separated by ≥72 hours.
  Arms: Combined Caffeine and L-Theanine (COM)
Dietary Supplement: Placebo — Participants receive placebo capsules filled with mannitol, a non-nutritive sugar alcohol with no known ergogenic or ergolytic effects. Capsules are identical in appearance, weight, and texture to the active supplement capsules and are taken orally with water 60 minutes before testing.
  Arms: Placebo (CON)

SUMMARY:
The aim of this clinical trial is to examine how caffeine and L-theanine, taken alone or together, affect both physical and cognitive performance in healthy, trained athletes. The study aims to answer whether these commonly consumed dietary ingredients can enhance strength, endurance, and hand-eye coordination under controlled laboratory conditions.

Researchers will compare four supplementation conditions:

Caffeine (CAF) - 3 mg per kilogram of body weight L-Theanine (THE) - 200 mg Combined Caffeine and L-Theanine (COM) - same doses together Placebo (CON) - mannitol (inactive substance) Each participant will complete all four test sessions in a randomized, double-blind, crossover design, with at least 72 hours between sessions. Capsules will be taken 60 minutes before testing to allow time for absorption. During each session, participants will perform a series of physical and cognitive tasks, including maximal isometric strength tests, an intermittent endurance test, and a computerized eye-hand coordination task.

The main hypothesis is that caffeine and L-theanine, alone or in combination, will improve strength and cognitive coordination compared with placebo. All participants are healthy competitive athletes between 18 and 30 years old. The study is conducted under standardized laboratory and indoor sports-hall conditions, with ethics approval obtained from the Sinop University Human Research Ethics Committee (Approval No. 2025/337).

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, crossover clinical trial investigates the acute effects of caffeine (CAF), L-theanine (THE), their combination (COM), and placebo (CON) supplementation on physical and cognitive performance in young, healthy, competitive athletes. Each participant completed all four experimental conditions in randomized order, separated by a minimum 72-hour washout period to minimize carryover effects. The randomization sequence was computer-generated by an independent researcher, and both participants and assessors were blinded to all conditions.

A total of 20 trained athletes (12 males, 8 females; 19.9 ± 2.4 years) participated. All were actively engaged in team or individual sports at a competitive level, with no history of cardiovascular, neurological, or musculoskeletal disorders, and no known intolerance to caffeine, theanine, or placebo components. Anthropometric and body composition data were collected using standardized procedures, including multi-frequency bioelectrical impedance analysis. Participants maintained normal caffeine consumption habits to preserve ecological validity and avoid withdrawal effects.

The supplementation protocol consisted of four conditions: (1) 3 mg/kg anhydrous caffeine, (2) 200 mg L-theanine, (3) a combination of both, and (4) placebo (mannitol). All supplements were encapsulated in visually identical gelatin capsules, and participants ingested five capsules with water 60 minutes before testing. Testing sessions were conducted at 09:00 a.m. to minimize circadian variability. Participants abstained from alcohol, strenuous exercise, and dietary supplements for 24 hours before each session, and replicated their pre-trial dietary intake based on 24-hour dietary logs.

All testing sessions were performed under standardized indoor laboratory conditions (22 ± 1 °C, 50 ± 5% humidity). The test sequence was fixed as eye-hand coordination, maximal isometric strength, and intermittent aerobic endurance, with adequate rest intervals between tests.

Primary outcomes included:

Maximal isometric strength, measured via handgrip, back, and leg dynamometry (Lafayette, Japan).

Intermittent aerobic endurance, assessed using the Yo-Yo Intermittent Endurance Test Level 1.

Eye-hand coordination, evaluated using a computerized test battery (EHC) that quantified accuracy, speed, and precision parameters.

A priori power analysis (f = 0.25, α = 0.05, 1-β = 0.80) determined a required sample size of 16 participants; 20 were recruited to allow for potential attrition. All 20 completed the study.

The study protocol was approved by the Sinop University Human Research Ethics Committee (Approval No. 2025/337), and written informed consent was obtained from all participants.

This trial aims to clarify whether acute ingestion of caffeine, L-theanine, or their combination exerts differential or synergistic effects on physical strength, endurance, and coordination in trained athletes, thereby contributing to the understanding of combined ergogenic aids in sports performance.

ELIGIBILITY:
Inclusion Criteria:

* Active participation in individual or team sports at a competitive level
* Age between [insert range, e.g., 18-30] years
* Absence of any known medical or metabolic disorder

Exclusion Criteria:

* History of cardiovascular, neurological, or musculoskeletal disorders within the past 12 months
* Known intolerance or hypersensitivity to caffeine or theanine
* Allergy to mannitol or other excipients used in capsule formulation
* Current use of prescription medications
* Physician-directed restriction of caffeine or theanine consumption.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Total Distance Covered in the Yo-Yo Intermittent Endurance Test Level 1 (meters) | 60 minutes post-supplement ingestion.
  Distance (m) completed during the Yo-Yo Intermittent Endurance Test Level 1 following standard protocol.
Peak Handgrip Force (kgf) | 60 minutes post-supplement ingestion.
  Highest handgrip force obtained from three maximal voluntary contractions using a calibrated digital dynamometer.
Peak Back Extension Force (kgf) | 60 minutes post-supplement ingestion.
  Highest value from three maximal voluntary contractions measured with a back strength dynamometer.
Peak Leg Extension Force (kgf) | 60 minutes post-supplement ingestion.
  Highest value from three maximal voluntary contractions measured using a leg dynamometer.
Eye-Hand Coordination Accuracy (EHC-A) | 60 minutes post-supplement ingestion.
  Accuracy percentage (%) obtained from the computerized eye-hand coordination test battery.
Eye-Hand Coordination Fast Speed Reaction Time (EHC-FS) | 60 minutes post-supplement ingestion.
  Reaction time (milliseconds) during the fast-speed EHC trial.
Eye-Hand Coordination Slow Speed Reaction Time (EHC-SS) | 60 minutes post-supplement ingestion.
  Reaction time (milliseconds) during the slow-speed EHC trial.
Eye-Hand Coordination Distance From Ball Center (EHC-DFBC) | 60 minutes post-supplement ingestion.
  Mean deviation from target center measured during coordination task.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinop University Facility, Sinop, Centarl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tuncer SY, Ozdenk S, Yildirim UC, Erkan D, Sari C, Gundem MC, Sar H, Yilmaz B, Karakulak I, Akca F. Acute effects of combined and isolated caffeine and theanine supplementation on physical and cognitive performance in competitive athletes: a randomized, double-blind, placebo-controlled crossover study. Front Nutr. 2026 Jan 26;12:1751673. doi: 10.3389/fnut.2025.1751673. eCollection 2025. PMID 41668720

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT07268573/Prot_SAP_000.pdf